CLINICAL TRIAL: NCT01296386
Title: An Open-label Phase 1 Study Assessing the Safety, Immunogenicity and Dose Response of IC84, a New Vaccine Against Clostridium Difficile, in Healthy Subjects
Brief Title: An Open-label Study Assessing Safety, Immunogenicity and Dose Response of IC84
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IC84-101
Record Dates: First submitted 2011-01-21; First posted 2011-02-15 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- IC84, 75 µg w/ Alum (Experimental): 75 µg w/ Alum (microgram with Alum)
  Interventions: Biological: IC84
- IC84, 75 µg w/o Alum (Experimental): 75 µg w/o Alum (microgram without Alum)
  Interventions: Biological: IC84
- IC84, 200 µg w/ Alum (Experimental): 200 µg w/ Alum (microgram with Alum)
  Interventions: Biological: IC84
- IC84, 200 µg w/o Alum (Experimental): 200 µg w/o Alum (microgram without Alum)
  Interventions: Biological: IC84

INTERVENTIONS:
Biological: IC84 — IC84, a recombinant fusion protein consisting of truncated Clostridium difficile (C. difficile) Toxin A and Toxin B, which will be administered at two different doses: 75 and 200 µg without or with Al(OH)3, respectively, intramuscular (i.m.) injection, four vaccinations on Day 0, 7, 28 and 56.

SUMMARY:
An open-label Phase 1 Study Assessing the Safety, Immunogenicity and Dose Response of IC84, A new vaccine against Clostridium Difficile (C. difficile), In healthy subjects

DETAILED DESCRIPTION:
This is an open-label, partially randomized, dose escalation Phase 1 study which will consist of a part A in healthy adults aged between ≥18 and <65 years and a part B in healthy elderly ≥65 years, the latter age group being the most vulnerable population to suffer from C. difficile infections.

Part A consists of 3 vaccinations on Day0, Day7 and Day21 with the following groups:

Group A: IC84 20 mcg (microgram)with Alum Group B: IC84 75 mcg (microgram)with Alum Group C: IC84 75 mcg (microgram)without Alum Group D: IC84 200 mcg(microgram)with Alum Group E: IC84 200 mcg(microgram)without Alum

Part A was already finished and part B is now ongoing. All information which could be find under the other sections are referring to the information on Part B.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults ≥18 years of age.
2. No clinically relevant pathological findings in any of the investigations at the Screening Visit including subjects with pharmacologically controlled conditions like hypercholesterolemia, hypertension, cardiovascular disease or non insulin-dependent diabetes mellitus. Minor deviations of laboratory values from the normal range may be accepted, if judged by the investigator to have no clinical relevance.
3. In female subjects, either childbearing potential terminated by surgery or 1 year post menopausal, or a negative serum pregnancy test during screening and the willingness not to become pregnant during the entire study period by practicing reliable methods of contraception.
4. Weight: ≥ 45.5 kg and <= 150 kg at Visit 0 (Screening Visit).
5. White blood cells ≥2,500/mm3 and <11,000/mm3 at Visit 0.
6. Platelets within normal limits at Visit 0.
7. Written informed consent obtained from the subject prior to any study related procedures.

Exclusion Criteria:

1. Use of any other investigational or non-registered medicinal product within 30 days prior to IC84 vaccination at Visit 1 (Day 0) and throughout the entire study period.
2. Active or passive vaccination four weeks before first vaccination at Visit 1 and during the entire study period.
3. Immunodeficiency including status post-organ-transplantation or immuno-suppressive therapy, and a family history of congenital or hereditary immunodeficiency.
4. Infection with the human immunodeficiency virus (HIV, a negative test result within 30 days before screening is acceptable), Hepatitis B virus (HBV, Hepatitis B surface antigen [HBsAg]) or Hepatitis C virus (HCV).
5. History of severe hypersensitivity reactions and anaphylaxis.
6. History of allergic bronchial asthma and severe allergic rhinoconjunctivitis.
7. Known hypersensitivity or allergic reactions to one of the components of the vaccine.
8. History of autoimmune disease, including Type I Diabetes mellitus. Subjects with vitiligo or thyroid disease taking thyroid hormone replacement are not excluded.
9. Any malignancy in the past 5 years. If treatment for cancer was successfully completed more than 5 years ago and the malignancy is considered to be cured, the subject may be enrolled.
10. Clinically significant hematological, renal, hepatic, pulmonary, central nervous, cardiovascular or gastrointestinal disorders, which are not adequately controlled by medical treatment within the last 12 weeks before IC84 vaccination at Visit 1 (Day 0) as judged by the site's Principal Investigator.
11. Systemic antibiotic use within four weeks prior to first vaccination and during treatment period (until Day 28).
12. Clinically significant diseases as judged by the investigator.
13. Administration of chronic (defined as longer than 14 days) immunosuppressants or other immune-modifying drugs within 30 days prior to IC84 vaccination at Visit 1 (Day 0) and during the study until Visit 5 (Day 28). (For corticosteroids this means prednisone or equivalent >= 0.05 mg/kg/day; topical and inhaled steroids are allowed.).
14. Periodic steroid injections, e.g., intra-articular, are not allowed within 30 days prior to first IC84 vaccination at Visit 1 (Day 0) and until Visit 5 (Day 28).
15. Intake of NSAID within three days prior to and within three days after all three vaccinations (Day 0, 7 and 21).
16. Acute febrile infections or exacerbation of chronic infection within four weeks prior to first vaccination at Visit 1 and during treatment period (until Day 21).
17. Body temperature > 37°C (oral) immediately prior to each vaccination.
18. Drug addiction within 6 months prior to Visit 0 [including alcohol dependence, i.e. more than approximately 60 g alcohol (approximately 1 liter of beer or 0.5 liter of wine) per day] indicated by an elevated MCV above normal value at the Screening Visit.
19. Inability or unwillingness to avoid more than the usual intake of alcohol [i.e., not more then 60 g alcohol (approximately 1 liter of beer or 0.5 liter of wine) per day] during the 48 hours after vaccination.
20. Pregnancy (positive pregnancy test during screening), lactation or unreliable contraception in female subjects with child-bearing potential ( and unreliable contraception in male subjects.
21. Not able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.
22. Blood donation within 4 weeks prior to first vaccination.
23. Clinically significant mental disorder not adequately controlled by medical treatment.
24. History of Guillain-Barré-Syndrome (GBS).
25. Any condition which might interfere with study objectives or would limit the subject's ability to complete the study in the opinion of the investigator.
26. Inability or unwillingness to provide informed consent.
27. Persons who are committed to an institution (by virtue of an order issued either by the judicial or the administrative authorities).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 82 (Actual)
Dates: Start 2010-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Rate of subjects with any SAE (Serious Adverse Event) possibly, probably or certainly related to the study vaccine at any time during the study | day 201
Rate of subjects with any unsolicited or solicited Grade 3 or higher adverse event possibly, probably or certainly related to the study vaccine at any time during the study | day 201
Rate of subjects with any unsolicited or solicited Grade 3 or higher adverse event possibly, probably or certainly related to the study vaccine during treatment phase (i.e. until Day 28) | day 201
Rate of subjects with solicited local AEs (Adverse Events) (injection site pain, tenderness, redness, swelling, induration, itching) within 1 week (Day 0-6) after each vaccination: Severity and duration. | 6 days after vaccination
Rate of subjects with solicited systemic AEs (headache, muscle pain, fever, flu-like symptoms, nausea, vomiting, rash, excessive fatigue) within 1 week (Day 0 6) after each vaccination: Severity and duration. | 6 days after vaccination
Rate of subjects with unsolicited non-serious AEs (including safety laboratory parameters (hematology, serum chemistry, urinalysis)) within 6 months after last vaccination: Severity and causality. | day 201
Rate of subjects with unsolicited non-serious AEs (including safety laboratory parameters (hematology, serum chemistry, urinalysis) during treatment phase (i.e., until Day 28): Severity and causality. | day 28

SECONDARY OUTCOMES:
Determination of vaccine (IC84) specific IgG levels on Day 0, 7, 14, 21, 28, 113 and 201 after the first vaccination using an Enzyme-Linked Immunosorbent Assay (ELISA) | day 201
Determination of C. difficile Toxin A- and Toxin B-specific IgG levels on Day 0, 7, 14, 21, 28, 113 and 201 after the first vaccination using an Enzyme-Linked Immunosorbent Assay (ELISA) | day 201
Determination of vaccine-induced C. difficile Toxin A- and Toxin B-neutralizing antibody levels on Day 0, 7, 14, 21, 28, 113 and 201 after the first vaccination using a Toxin Neutralization Assay (TNA) | day 201

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Ayad, Dr., Study Chair — Valneva Austria GmbH
Locations (3):
- Austria (2):
  - Privatklinik Leech, Graz
  - Medizinische Universität Wien, Vienna
- St. Imre Teaching Hospital, Budapest, Hungary

REFERENCES:
- [Derived] Bezay N, Ayad A, Dubischar K, Firbas C, Hochreiter R, Kiermayr S, Kiss I, Pinl F, Jilma B, Westritschnig K. Safety, immunogenicity and dose response of VLA84, a new vaccine candidate against Clostridium difficile, in healthy volunteers. Vaccine. 2016 May 17;34(23):2585-92. doi: 10.1016/j.vaccine.2016.03.098. Epub 2016 Apr 11. PMID 27079932